CLINICAL TRIAL: NCT03357718
Title: Oral Dexmedetomidine vs Midazoam For Premedication And Emergence Delirium in Children Undergoing Dental Treatment
Brief Title: Oral Dexmedetomidine vs Midazoam For Premedication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sultan KELES, Assist. Prof.Dr., Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017/18
Record Dates: First submitted 2017-11-24; First posted 2017-11-30 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2017-11

CONDITIONS: Premedication
Keywords: premedication
MeSH Terms: interventions — Dexmedetomidine; Midazolam

STUDY DESIGN:
Intervention Model Description: Retrospective clinical trial
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): 2 µg/kg Precedex
  Interventions: Drug: Precedex
- Midazolam (Active Comparator): 0.5 mg/kg dormicum
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Precedex — 2 µg/kg oral
  Other Names: Dexmedetomidine
  Arms: Dexmedetomidine
Drug: Midazolam — 0.5 mg/kg
  Other Names: Dormicum
  Arms: Midazolam

SUMMARY:
The aim of this study was to compare the effect of 2 µg/kg of oral dexmedetomidine (DEX) and 0.5 mg/kg dormicum as premedication among children undergoing dental procedures.

DETAILED DESCRIPTION:
The study involved 52 children between 3-7 years of age, ASA I , who underwent full-mouth dental rehabilitation. The DEX group (n=26) received 2 µg/kg DEX in apple juice, and the control group (n=26) received 0.5 mg/kg midazolam in apple juice.

The patients' scores on the Ramsey sedation scale (RSS), parental separation anxiety scale, mask acceptance scale, post-anesthesia emergence delirium scale (PAEDS), and hemodynamic parameters were recorded. The data were analyzed using chi-square test, Fisher's exact test, student t test, and analysis of variance in SPSS.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria is age between 3 to 7 years and American Society og Anesthesiology (ASA) grade 1.

Exclusion Criteria:

* The exclusion criteria included congenital disease, DEX, propofol allergy, asthma, mental retardation and those children parents refuse to participate study.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-05-30 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Ramsey Sedation Scale | 45 minutes after premedication
  Sedation level is evaluated due to patient behavior. 1= Patient is anxious and agitated or restless or both, 2=Patient is cooperative, oriented, and tranquil, 3=Patient responds to command only, 4=Patient exhibits brisk response to light glabellar tap, 5=Patient exhibits sluggish response to light glabellar tap, 6=Patient exhibits no response.A Ramsay sedation score '1' was considered as unsatisfactory and "≥ 2" was considered as satisfactory sedation.

SECONDARY OUTCOMES:
Parental Separation Anxiety Scale | Preoperative
  Behavior of the child on seperation from the parents was assessed according to a four-point scale, i.e., the parental seperation anxiety scale (PSAS): 1= Easy seperation, 2=Whimpers but easily reassured, 3=Cries and cannot be easily reassured, but not clinging to parents, 4=Cries and clinging to parents. A PSAS score of 1 and 2 were considered as 'successful parental seperation'.
Mask Acceptance Score | Before induction
  Mask acceptance was evaluated using a four-point scale, i.e., mask acceptance scale (MAS):
  1=Excellent (unafraid, cooperative, and accepts mask easily), 2=Good (slight fear of mask , easily reassured), 3=Fair (moderate fear of mask, not calmed with reassurance), 4=Poor (terrified, crying, or combative). The score of 1 and 2 considered as 'satisfactory' mask acceptance.

CONTACTS AND LOCATIONS:
Overall Officials: Sultan KELES, Dr., Principal Investigator — Adnan Menderes University Faculty of Dentistry Aydın

IPD SHARING:
Plan to Share IPD: No
Results

REFERENCES:
- [Background] Kumari S, Agrawal N, Usha G, Talwar V, Gupta P. Comparison of Oral Clonidine, Oral Dexmedetomidine, and Oral Midazolam for Premedication in Pediatric Patients Undergoing Elective Surgery. Anesth Essays Res. 2017 Jan-Mar;11(1):185-191. doi: 10.4103/0259-1162.194586. PMID 28298782